CLINICAL TRIAL: NCT04475484
Title: Online Survey on Psychological Impact of COVID-19 Epidemic on School-age Children
Acronym: PSICOcs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: PSICOcs_2020
Record Dates: First submitted 2020-07-06; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Investigating Psychological Impact; Confinement Measures; Coronavirus Outbreak; School-age Children
Keywords: coronavirus epidemic; Children; Schooling

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- School-age children: School-age children from primary school to high school (about age 6 to 18) in the Academy of Lyon
  Interventions: Other: Online questionnaire

INTERVENTIONS:
Other: Online questionnaire — Parents will receive a link to an online questionnaire through computing services of Lyon's Academy. They have to give their consent to allow their child to participate in the study. Then, children can complete the online questionnaire.
  The questionnaire starts with few explanations on the context of the study, and ends with psycho-education advices and what to do in the event of psychological distress.

SUMMARY:
The coronavirus outbreak is a stressful event for the whole population. Confinement measures are protective against the risk of dissemination of the virus, but they can also lead to several psychological symptoms. In children, a study in China has reported about 20% of depressive or anxious troubles in school-age children after a 4-week period of confinement.

In France, confinement lasted about 8 weeks. School resumed on May 11th for primary school children and on June 2nd for secondary school children.

In this survey, we aim at exploring the psychological status of these children and the impact on their schooling, for better understanding, support and prevention. Through this online questionnaire, we also aim at giving some psycho-education advices. Finally, we could identify some subgroups of children particularly vulnerable, and organise some specific support for them in coming months.

ELIGIBILITY:
Inclusion Criteria:

* school-age children in the Academy of Lyon
* parental consent

Exclusion Criteria:

-

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: School-age children from primary school to high school (about age 6 to 18) in the Academy of Lyon
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of children presenting signs of psychological suffering during confinement. | We plan to address a first online questionnaire in June 2020 (school resumption after confinement), and a follow-up questionnaire 3 months later, in September 2020.
  We plan to assess the psychological status of children during coronavirus outbreak : negative and positive feeling during confinement, worries and expectations about school resumption.
  We also aim at correlating high stress levels with environmental or/and temperamental factors.

CONTACTS AND LOCATIONS:
Locations (1):
- hôpital Femme Mère Enfant, Bron, France